CLINICAL TRIAL: NCT04755634
Title: Shafer Width and Girth: The Use of Injectable Fillers for Penile Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shafer Clinic Fifth Avenue (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00034295
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Micropenis
MeSH Terms: conditions — Penis agenesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): This is a prospective, single-arm, single-center study
  Interventions: Device: Hyaluronic Acid

INTERVENTIONS:
Device: Hyaluronic Acid — Injectable

SUMMARY:
Injectable filler will be performed by Principal Investigator under sterile conditions for the enhancement of girth and surface area of the penis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males,
* 21 to 65 years of age,
* Seeking enhancement of their penile width and girth.

Exclusion Criteria:

* Patient with a history of psychological or psychiatric illness,
* Congenital or acquired penile malformation,
* Previous plastic surgery or non-invasive treatments of their penis,
* Any chronic disease such as vascular disorder, urological disorder, myocardial infarction, hypertension, cerebrovascular accident or coagulopathy.
* Patients with a history of allergic reactions to hyaluronic acid derivatives
* Individuals with penises measured less than 6 cm in length in the flaccid position
* Individuals with penises greater than 12.5 cm in length in the flaccid position.
* Individuals with uncircumcised penises

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Increase in penile width and girth | 1 year
  Three-dimensional (3D) surface images taken by a digital stereophotogrammetry system at the baseline will be compared to the images taken at 1 year post-treatment follow up.

SECONDARY OUTCOMES:
Duration of increase in penile width and girth | 1 year
  For how long duration the treatment will produce a measurable difference in penile size.

CONTACTS AND LOCATIONS:
Overall Officials: David Shafer, MD, Principal Investigator — Shafer Clinic Fifth Avenue
Locations (1):
- Shafer Clinic Fifth Avenue, New York, New York, United States